CLINICAL TRIAL: NCT00307814
Title: A Randomized, Open-Label Clinical Evaluation of PROCRIT (Epoetin Alfa) for Maintenance Phase Treatment of Patients With Anemia Due to Chronic Kidney Disease
Brief Title: A Study to Evaluate PROCRIT (Epoetin Alfa) for Maintenance Phase Treatment of Patients With Anemia Due to Chronic Kidney Disease (PROMPT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005101
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Chronic Renal Insufficiency
Keywords: Anemia; Low Blood Count; Chronic Kidney Failure; Chronic Kidney Disease; epoetin alfa; recombinant human erythropoietin
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of less frequent dosing of PROCRIT (Epoetin alfa) in patients with anemia due to Chronic Kidney Disease (CKD) as assessed by hemoglobin maintenance, adverse events and health-related quality of life.

DETAILED DESCRIPTION:
Epoetin alfa has been widely utilized as treatment for anemia associated with Chronic Kidney Disease (CKD). Epoetin alfa has been shown to increase hemoglobin (Hb) levels by an average of 1.5 g/dL to 2 g/dL in these patients over 12 weeks (Data on file Ortho Biotech Products, L.P.). This improvement in Hb levels is maintained while the patient is receiving Epoetin alfa and is associated with significant improvements in survival, exercise tolerance, and quality of life. Literature has suggested that epoetin alfa can be given less frequently and still maintain an optimal hemoglobin while also allowing patient's greater convenience. This study will further confirm that less frequent dosing of epoetin alfa is safe and effective. This is an open-label, randomized multicenter study in patients with CKD. CKD patients who are currently receiving PROCRIT therapy for at least 2 months or more and with a stable Hb (>= 11g/dL) will be randomized to one of four treatment groups. A stable Hemoglobin will be defined as a value that is ± 10% for 3 consecutive laboratory values.

This study is designed to demonstrate that there is no meaningful difference in hemoglobin level with more extended dosing regimens as compared to once weekly. A clinically meaningful difference is defined as a difference that is less than 10%. Patients will be randomized to one of 4 treatment groups: All will receive subcutaneous (under the skin) Epoetin alfa for a period of 16 weeks.

Group 1: 10,000 units every week Group 2: 20,000 units every two weeks Group 3: 30,000 units every three weeks Group 4: 40,000 units every four weeks

ELIGIBILITY:
Inclusion Criteria:

* CKD patients (defined as serum creatinine 1.5 to 6.0 mg/dL for women and 2.0 to 6.0 g/mg/dL for men)
* Stable Hb (>= 11.0g/dL) and currently receiving PROCRIT therapy for 2 months or more. A stable Hemoglobin will be defined as a value that is ± 10% for 3 consecutive laboratory values.

Exclusion Criteria:

* Lactating or pregnant women
* Uncontrolled hypertension
* Known hypersensitivity to mammalian cell-derived products and human albumin
* Receiving dialysis or scheduled to receive dialysis during the course of the study
* gastrointestinal bleeding
* Severe Congestive Heart Failure (New York Heart Association Class IV)
* Concurrent chemotherapy for cancer
* History of/or active blood disorders, liver diseases or seizures
* HIV positive
* Received a kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2002-01; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is hemoglobin maintenance. Also, patients will be assessed for incidence and severity of adverse events and vital signs (blood pressure) during the 16 week study period.

SECONDARY OUTCOMES:
The secondary variable is Quality of Life and Hemoglobin Change over Time

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Result] Provenzano R, Bhaduri S, Singh AK; PROMPT Study Group. Extended epoetin alfa dosing as maintenance treatment for the anemia of chronic kidney disease: the PROMPT study. Clin Nephrol. 2005 Aug;64(2):113-23. doi: 10.5414/cnp64113. PMID 16114787
- See also: A Randomized, Open-label Clinical Evaluation of PROCRIT (Epoetin ala) for Maintenance Phase Treatment of Patients with Anemia due to Chronic Kidney Disease (PROMPT Study) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=926&filename=CR005101_CSR.pdf